CLINICAL TRIAL: NCT03273426
Title: Prediction of Pathologic Complete Response by Multiple Core Needle Biopsy or Vacuum Assisted Biopsy Before Surgery in Breast Cancer With Complete Clinical Response After Neoadjuvant Chemotherapy.
Brief Title: Prediction of pCR by Preoperative Biopsy in Breast Cancer With cCR After Neoadjuvant Chemotherapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wonshik Han, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUHBCC002
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Needle

STUDY DESIGN:
Intervention Model Description: Comparison of pathological findings for residual tumor between minimally-invasive biopsy procedure and subsequent wide excision of the biopsied area
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Core needle Biopsy (Experimental): Ultrasound-guided core needle biopsy (14G, ≥5 cores recommended) for complete clinical response (cCR) or near-cCR predicted by MRI.
  Interventions: Procedure: Minimally-invasive biopsy; Procedure: wide excision
- Vacuum-assisted biopsy (Experimental): Vacuum-assisted biopsy (10G, ≥5 cores recommended) for complete clinical response (cCR) or near-cCR predicted by MRI.
  Interventions: Procedure: Minimally-invasive biopsy; Procedure: wide excision

INTERVENTIONS:
Procedure: Minimally-invasive biopsy — Intervention (core needle biopsy (14G) or vacuum-assisted biopsy(10G)) for complete clinical response (cCR) or near-cCR predicted by MRI.
  Other Names: vacuum-assisted biopsy; core-needle biopsy
Procedure: wide excision — Surgical wide excision of the biopsied area.

SUMMARY:
The purpose of this study is to evaluate the ability of preoperative biopsy to predict correctly pathologic complete response in breast cancer patients with complete clinical response after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Breast cancer patients who received neoadjuvant chemotherapy and is predicted to have achieved pathologic complete response (pCR) on MRI will enrolled. The enrolled patients will undergo either US-guided multiple core needle biopsy or US-guided vacuum-assisted biopsy of the tumor bed where it had been marked with an indicator (clip). The patient will undergo subsequent wide excision of the tumor bed. Histopathologic findings of the biopsy and the surgical specimen will be compared for pCR, and the ability of preoperative biopsies to predict pCR will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients

* with unilateral primary cancer pathologically confirmed before neoadjuvant chemotherapy (NAC)
* who received NAC
* with detectable lesion / clip marker on ultrasound
* with cT1-T3 tumors
* clinical and imaging complete or near-complete response on MRI
* with informed consent

Exclusion Criteria:

* Multifocal cancer
* Residual microcalcification
* Contralateral breast cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wonshik Han, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
IPD including study protocol, informed consent form, clinical study report and analytic code will be shared.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication.
Access Criteria: PI will review requests for IPD.

REFERENCES:
- [Derived] Pfob A, Sidey-Gibbons C, Lee HB, Tasoulis MK, Koelbel V, Golatta M, Rauch GM, Smith BD, Valero V, Han W, MacNeill F, Weber WP, Rauch G, Kuerer HM, Heil J. Identification of breast cancer patients with pathologic complete response in the breast after neoadjuvant systemic treatment by an intelligent vacuum-assisted biopsy. Eur J Cancer. 2021 Jan;143:134-146. doi: 10.1016/j.ejca.2020.11.006. Epub 2020 Dec 8. PMID 33307491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sep 2016 to Feb 2018 at Breast Care Center, Seoul National University Hospital
Pre-assignment Details: All enrolled patients completed the protocol for minimally-invasive biopsy and subsequent wide excision.
Groups:
- Core Needle Biopsy: Image-guided core needle biopsy (14G, ≥5 cores recommeded) for complete clinical response (cCR) or near-cCR predicted by MRI.
  The patients were assigned to either core needle biopsy or vacuum-assisted biopsy alternatively.
- Vacuum-assisted Biopsy: Image-guided vacuum-assisted biopsy (14G, ≥5 cores recommeded) for complete clinical response (cCR) or near-cCR predicted by MRI.
  The patients were assigned to either core needle biopsy or vacuum-assisted biopsy alternatively.
Period: Overall Study
Arm/Group | Core Needle Biopsy | Vacuum-assisted Biopsy
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Needle Biopsy | Vacuum-assisted Biopsy | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Standard Deviation); unit: years] | 52 (10.74) | 46.5 (10.03) | 49 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 20 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 20 | 20 | 40
Tumor size before neoadjuvant chemotherapy [Mean (Standard Deviation); unit: millimeters] — Maximum tumor size on imaging in mm before neoadjuvant chemotherapy
  millimeters | 29.55 (15.51) | 31.8 (12.90) | 30.68 (14.13)

OUTCOME MEASURES:

1. Primary Outcome: Negative Predictive Value
Description: Percentage of participants with pathologic complete response (pCR) confirmed by surgical excision in patients predicted by biopsy to have pCR
Time Frame: 2 weeks
Population: Number of participants with no tumor on biopsy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: Ultrasound-guided core needle biopsy + vacuum-assisted biopsy
Arm/Group | Core Needle Biopsy | Vacuum-assisted Biopsy | Total
Number analyzed (Participants) | 17 | 14 | 31
percentage of participants | 88.2 [71.94 to 95.64] | 85.7 [64.37 to 95.22] | 87.1 [74.92 to 93.85]

2. Secondary Outcome: False Negative Rate
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Core Needle Biopsy | Vacuum-assisted Biopsy
Number analyzed (Participants) | 20 | 20
percentage of participants | 40 | 25

ADVERSE EVENTS:
Time Frame: 2 weeks after intervention (CNB or VAB)
Arm/Group | Core Needle Biopsy | Vacuum-assisted Biopsy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Needle Biopsy (N=20) | Vacuum-assisted Biopsy (N=20)
bleeding (Surgical and medical procedures) | 0 (0) | 1 (1) — post-biopsy bleeding
hematoma (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03273426/Prot_SAP_000.pdf
  • Informed Consent Form (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03273426/ICF_001.pdf